CLINICAL TRIAL: NCT07350772
Title: Atypical Lupus Presentations and Their Prognostic Implications
Brief Title: It is an Observational Study That Compare Prognosis of Typical and Atypical Systemic Lupus Erythematosus Presentation
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmin Abdelfattah Mohamed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med--25-12-7MD
Record Dates: First submitted 2025-12-27; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systemic lupus erythematosus patients with typical presentations
- Systemic lupus erythematosus patients with atypical presentations

SUMMARY:
Atypical presentations of SLE including unusual initial symptoms, predominant organ involvement, late-onset disease and ANA-negative remain poorly characterized. These forms are often associated with delayed diagnosis and potentially worse clinical outcomes. Most existing studies focus on isolated rare manifestations rather than analyzing atypical SLE as a cohesive category. Understanding these differences is crucial and this study aims to compare atypical and typical SLE presentations to clarify variations in prognosis, treatment requirements and subsequent organ involvement.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as SLE according toSLICC 2012Classification Criteria[13] :

A. Patients presented with typical lupus presentation:

1. age of onset (20-50)
2. common initial manifestations as constitutional manifestations,arthritis, mucocutaneousmanifestationslike malar rash, photosensitivity and hair falling.
3. patients with ANA positive.

B. Patients presented with atypical lupus presentation:

1. any clinical presentation not belonging to classic common SLE onset features, including but not limited to:

   * Neuropsychiatric onset: seizure, psychosis, aseptic meningitis, transverse myelitis
   * Cardiopulmonary onset: pulmonary hypertension, acute pneumonitis, myocarditis, pulmonary hemorrhage
   * Gastrointestinal onset: mesenteric vasculitis, intestinal pseudo obstruction, pancreatitis
   * Hematologic severe onset: isolated severe thrombocytopenia, autoimmune hemolytic anemia, thrombotic microangiopathy
   * Dermatologic atypical onset: bullous lupus, panniculitis, vasculitic ulcers
   * Myositis
   * Fever of unknown origin (FUO) as sole initial presentation
   * Thrombotic events
   * Generalized lymphadenopathy.
2. Patients with dominant organ affection.
3. patients with late onset SLE.
4. patients with ANA negative SLE. C.Patients who can provide informed consent.

exclusion criteria:

1. Patients whose initial symptoms are clearly attributable to infection, sepsis or another non-SLE condition.
2. Patients with chronic pre-existing diseases that may mimic or obscure the initial SLE presentation (e.g. primary epilepsy, primary pulmonary hypertension, chronic liver or GI disease).
3. Patients in whom onset features cannot be reliably classified as typical or atypical due to mixed or unclear presentation.

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 400 patients diagnosed according to SLICC classification criteria as systemic lupus erythematosus[13] including 3oo patients with typical common SLE presentation and 100 patients with atypical presentation as rare manifestations,ANA negative lupus, late onset lupus.Patients will be collected from Rheumatology outpatient clinic - Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Disease activity measured by SLEDAI-2K score | Baseline (0 month), 6 months, 12 months
  SLEDAI-2K score will be calculated for each participant. Data will be reported as mean ± SD and compared between patients with typical and atypical SLE presentations
Organ damage accrual measured by SDI score | 6 months, 12 months
  Systemic Lupus International Collaborating Clinics Damage Index (SDI) will be assessed to evaluate irreversible organ damage. Data will be reported as mean ± SD and compared between patients with typical and atypical SLE presentations

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals,sohag ,sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07350772/Prot_SAP_000.pdf